CLINICAL TRIAL: NCT06883812
Title: Continuous Glucose Monitoring in Prediabetes With Health Education Videos
Acronym: G2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David S Black, PhD (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor-Investigator, David S Black, PhD, Tenured Associate Professor of Population and Public Health Sciences, University of Southern California
Organization: University of Southern California (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UP-23-01001(a); 3P50MD017344-03S3 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes
Keywords: Prediabetes; Glucose control; Feedback; Health education; Artificial intelligence; Behavioral analysis
MeSH Terms: conditions — Prediabetic State; Health Education

STUDY DESIGN:
Intervention Model Description: An AB sequential condition design with CGM automated continuous glucose recording with glucose level masked and unmasked phases.
Masking Description: Participants are blinded to glucose values during Phase A. The CGM system generates automated records of glucose and does not require observation from an outcomes assessor. The investigator does not engage with participants and becomes aware of unmasking after trial is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Group (Other): Participants wear a CGM on the back of the arm. During Phase A, glucose values are not visible to participants. During Phase B, glucose values are visible via the phone app.
  Interventions: Device: CGM

INTERVENTIONS:
Device: CGM — The CGM sensor is worn on the back of the arm and glucose levels are recorded continuously but levels are not shown on the participant's phone app in phase A.

SUMMARY:
The objective of this project is to deliver a behavior health education video series that combines wearable continuous glucose monitoring (CGM) with smartphone feedback and video clips generated by artificial intelligence (AI) software to improve glycemic control among individuals with prediabetes. The goal is to prevent transition to type 2 diabetes and advanced metabolic complications.

DETAILED DESCRIPTION:
A health education video series, ¡Mi Control!, led by community health workers known as Promotores de Salud (PdS), will be integrated with continuous glucose monitoring (CGM) to support self-monitoring of glucose levels and excursions. Study G2 is a Phase 0 feasibility study enrolling 30 Spanish- and/or English-speaking PdS who test positive for prediabetes via a finger-prick A1c% screening. Participants will wear CGM devices for 20 days, with glucose data masked for the first 10 days and unmasked for the next 10 days. During the unmasked phase, participants will receive daily health education videos on their smartphones. The study will compare the duration of glucose excursions between the masked and unmasked phases to assess the impact of CGM feedback and health education on glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes by finger prick blood A1C%
* Centers for Disease Control and Prevention (CDC) prediabetes risk test score of 5 or higher
* Willingness to wear CGM sensor
* Community health worker

Exclusion Criteria:

* Currently pregnant
* Less than 18 years of age, which is adult in California
* Diagnosed with any disorder that interferes with glucose
* Influential medical disorder/event affecting ability to participate in study
* Incompatible smartphone device not pairing with Dexcom G6 app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Glucose levels | Maximum of 20 days of continuous wear
  Mean glucose in mg/dL

SECONDARY OUTCOMES:
Time out of range > 140 mg/dL (TOR) | Maximum of 20 days of continuous wear
  Time out of range > 140 mg/dL (TOR)

CONTACTS AND LOCATIONS:
Overall Officials: David S Black, PhD MPH, Principal Investigator — University of Southern California Keck School of Medicine
Locations (1):
- Southern California Center for Latino Health SCCLH, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing is set up with affiliate USC-CHLA P50 Center universities and hospitals under a registered data use agreement (DUA). Data and protocol documentation will be posted on the Open Science Framework
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: No longer than one year after the completion of the trial. Researchers can obtain de-identified data and statistical codes after publication of the study outcomes by email request and as supplemental material in future journal publications.
Access Criteria: Publicly available link or by request to PI or directly obtained as supplemental material from the website of the journal publication.
URL: https://www.clinicaltrials.gov

REFERENCES:
- See also: Dexcom G CGM system specifications — https://www.dexcom.com